CLINICAL TRIAL: NCT05861154
Title: Effectiveness of Laser Photobiomodulation Therapy in Reducing Child Pain During Local Anesthesia Injection (a Randomized Controlled Clinical Trial)
Brief Title: Effectiveness of Laser Photobiomodulation Therapy in Reducing Child Pain During Local Anesthesia Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aliaa Hamouda (Other)
Responsible Party: Sponsor-Investigator, Aliaa Hamouda, Assistant Lecturer of Pediatric Dentistry, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: #11
Record Dates: First submitted 2023-04-28; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Local Anesthesia Injection Pain
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation (Experimental)
  Interventions: Device: Photobiomodulation
- Topical anesthesia (Active Comparator)
  Interventions: Drug: Benzocaine Gel

INTERVENTIONS:
Device: Photobiomodulation — A diode laser (Sirolaser blue laser system, Sirona Dental Systems GmbH, Fabrikstraße 31, 64625 Bensheim, Germany) of Wavelength 660 nm will be used and the laser parameters will be set as follows: Power 0.1 W, energy 6 J, Continuous wave, Irradiation time 60 Seconds; energy Tip area 0.5 cm2, fluence 12 J/cm2 will be applied at the site of needle penetration.
  It should be noted that before each application, the output of the laser device will be checked using the aiming beam on flat surface; both the patient and the operator will wear safety goggles during the irradiation.
  Arms: Photobiomodulation
Drug: Benzocaine Gel — a 20% Benzocaine topical anaesthetic gel will be applied. To increase the absorption of the topical anaesthetic gel, soft tissues will be dried with (2 x 2 cm) gauze. Topical anaesthetic gel will be applied at the site of needle penetration and left in contact with the soft tissues for one minute in order to to maximize its effect.
  Arms: Topical anesthesia

SUMMARY:
This study aimed to evaluate the impact of laser photobiomodulation therapy used as pre-anesthetic technique to reduce child pain during local anesthesia administration

ELIGIBILITY:
Inclusion Criteria:

* Completion of the written informed consent form by parents/guardian.
* Children with dental behavior score of 3 or 4 according to the Frankel behavior rating scale.
* Patients whom their maxillary primary molars are indicated for pulpotomy and SSC restoration.
* Lack of history of allergy to the materials used for anesthesia and sulfite
* Children free of any systemic disease or special health care needs (ASA 1)

Exclusion Criteria:

* Children who receive any analgesic drugs at least 24 hours before treatment.
* Any inflammation or lesion in the injection site
* Patients who have previous bad experience of dentistry were excluded to eliminate the possible impact of the child's previous painful or stressful experiences
* Child coming for emergency treatment of pain

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | during local anesthesia administration
  A brief demonstration of the pulse oximeter will be performed, and the patient will be instructed to remain still and avoid hand movement in order to obtain accurate readings. The pulse oximeter will be placed on the patient's index finger to measure the baseline heart rate (prior to administering the LA), and another measurement will be taken during the LA administration. Heart rate will be recorded at 2-minute intervals and the mean heart rate measurement will be calculated.
Pain Reaction | during local anesthesia administration
  The Sound, Eye, Motor (SEM) Scale will be used to assess pain. It encompasses the following parameters: (1) Sound, (2) Eye and (3) Motor. The sounds, eye symptoms and body movements of each child will be independently evaluated by a blind impartial observer using the recorded video tapes. The slightest manifestation of the patient's sound, eyes, or motion is graded in four levels: comfort, mild, moderate, and severe discomfort, and subsequently given grades 1, 2, 3, 4, respectively. The SEM score will be calculated by adding the three parameter grades.
Perceived Pain | immediately after local anesthesia administration
  To subjectively record pain during LA injection, a modified face scale will be used. It comprises three schematic faces with different facial expressions for happy and sad faces representing: (A) satisfaction; (B) indifference; and (C) dissatisfaction, respectively. Each child will be taught before injection how to use the scale by modelling and then asking each participant to recall the last time she or he felt something painful and select the facial expression that best represented his or her experience of discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Hamouda, MSc, Principal Investigator — Alexandria University; Amani Khalil, PhD, Study Chair — Alexandria University; Laila El-Habashy, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Hamouda AA, El-Habashy LM, Khalil A. The use of laser photobiomodulation as pre-anesthetic tissue management technique in reducing injection pain in children. BMC Oral Health. 2024 Jun 22;24(1):717. doi: 10.1186/s12903-024-04430-3. PMID 38909229